CLINICAL TRIAL: NCT02214732
Title: A Randomized Controlled Trial of Mindfulness Based Cognitive Therapy for Psychological Distress in Pregnancy
Brief Title: Mindfulness Based Cognitive Therapy for Psychological Distress in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Centre for Child, Family & Community Research (Other); Alberta Family Wellness Initiative (Unknown)
Responsible Party: Principal Investigator, Lianne Tomfohr-Madsen, Assistant Professor of Psychology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB13-0860
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Depression; Anxiety; Stress
Keywords: Pregnancy; Postpartum; Mindfulness Based Cognitive Therapy; Depression; Anxiety; Stress; MBCT; Actigraphy
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCT + Treatment as Usual (TAU) (Experimental): Behavioural: Mindfulness Based Cognitive Therapy
  Participants in the MBCT group attend an 8 week course of a modified MBCT program for pregnant women, delivered by a licensed clinical psychologist.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment as Usual (TAU) (No Intervention): Participants in the TAU group access community resources for pregnant women experiencing psychological distress.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — The modified MBCT program for pregnant women is an 8-session group intervention that aims to help women change their relationship to the thoughts, feelings, and bodily sensations that can lead to psychological distress. Participants are guided to recognize and disengage from unhelpful mind states characterized by self-perpetuating patterns of ruminative thought. The intervention was modified to address pregnant women's physical and emotional needs, as well as their risk of perinatal mood episodes.
  Other Names: MBCT
  Arms: MBCT + Treatment as Usual (TAU)

SUMMARY:
Anxiety, stress and depression are common during pregnancy and in the postpartum period. The lack of empirically supported, non-pharmaceutical interventions for psychological distress in pregnancy is a significant gap in the literature, especially given many pregnant women's preference for non-pharmaceutical treatments. This study will evaluate the efficacy of Mindfulness Based Cognitive Therapy (MBCT) program in reducing measures of psychological distress (e.g., symptoms of stress, depression and anxiety) in a group of pregnant women endorsing high levels of distress.

ELIGIBILITY:
Inclusion Criteria:

Eligible women for this study

* are between 12 and 28 weeks of gestation,
* are experiencing psychological distress (elevated perinatal anxiety, mild depressive symptoms, or high-levels of self-reported stress)

Exclusion Criteria:

* current suicidality
* current substance abuse or dependence
* experience a current major depressive episode
* have been diagnosed with bipolar disorder or other disorders that have a psychotic, dissociative, hallucinatory, or delusional component
* taking prescribed medications that affect sleep or mood

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Edinburgh Postpartum Depression Scale scores from baseline to 3 months follow-up postpartum | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum (3 months after the birth of a person's baby)
  Symptoms of depression will be assessed using the 10-item, self-report Edinburgh Postpartum Depression Scale (EPDS). The EPDS has been validated against interview schedules and other self-report instruments.

SECONDARY OUTCOMES:
Change in Pregnancy Related Anxiety Measure scores from baseline to post-treatment | Baseline (Week 1), Post-Treatment (Week 10)
  The Pregnancy Anxiety Measure, a 10-item instrument will be used to examine the extent to which women are worried about their own and baby's health, labour, delivery and caring their new baby.
Change in Perceived Stress Scale (PSS-10) scores from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  This questionnaire will be used in assessing the perception of stress. The questions are in regards to participant's feelings and thoughts during the previous month. It was designed to be used in community samples. The items are assessing perceived helplessness and self-efficacy.
Change in Pittsburgh Sleep Quality Index (PSQI) scores from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  The PSQI instrument will be used in assessing participant's sleep quality. There are seven components of the PSQI and these are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction.
Change in objective measures of sleep using Wrist Actigraphy from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  Actigraphy monitoring provides objective information on circadian rhythm amplitude, acrophase, as well as indices of sleep efficiency, sleep latency, total sleep time, and number and frequency of awakenings. The use of actigraphy has been demonstrated sensitive to treatment effects, while being less costly and intrusive than polysomnography.
Change in salivary cortisol profile from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  All samples are assayed for salivary cortisol using a highly sensitive enzyme immunoassay.
Change in measures of blood pressure (BP) from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  BP data will be collected using an automatic, calibrated, oscillometric BP monitor and a BP cuff on the upper part of the dominant arm.
Changes in measures of heart rate variability from baseline to 3 months | Baseline (Week 1), Post-Treatment (Week 10), 3 months follow-up postpartum
  Measures of heart rate (bpm) will be recorded noninvasively using a HIC-2000 Bio-electric Impedance Cardiograph and the Cardiac Output Program, developed by Bio-Impedance Technology.

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Riley Park Maternity Clinic, Calgary, Alberta
  - University Of Calgary, Calgary, Alberta

REFERENCES:
- [Derived] Tomfohr-Madsen LM, Campbell TS, Giesbrecht GF, Letourneau NL, Carlson LE, Madsen JW, Dimidjian S. Mindfulness-based cognitive therapy for psychological distress in pregnancy: study protocol for a randomized controlled trial. Trials. 2016 Oct 13;17(1):498. doi: 10.1186/s13063-016-1601-0. PMID 27737714